CLINICAL TRIAL: NCT04201015
Title: Mechanisms, Safety and Efficacy of Optimising Pacemaker Heart Rate for Contractility: Effects on Walk Time, Cardiac Remodelling and Quality of Life
Brief Title: Optimising Pacing for Contractility 2
Acronym: OPT-cont 2
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Klaus K Witte, MD, Prinicipal Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 277578
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure, Systolic; Pacemaker
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the technician doing the programming will know how the pacemaker has been set.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard rate-response settings (No Intervention): Patients allocated to standard rate-response settings.
- Rate-response settings off (Active Comparator): Patients allocated to deactivated rate-response settings.
  Interventions: Device: Heart rate optimisation using force frequency data
- Optimized rate-response settings (Experimental): Patients allocated to optimised rate-response settings.
  Interventions: Device: Heart rate optimisation using force frequency data

INTERVENTIONS:
Device: Heart rate optimisation using force frequency data — Programming heart rate rise according to the force frequency relationship
  Arms: Optimized rate-response settings; Rate-response settings off

SUMMARY:
The investigators have demonstrated that they can reliably identify an optimum heart rate range for contractility of the left ventricle in patients with chronic heart failure (CHF). They have also demonstrated in an acute cross-over and a small parallel group feasibility study that keeping the heart rate in this range (versus standard rate-response programming) in patients with CHF is associated with increased exercise time on a treadmill (around 60s or 10%). They now want to explore in a randomised, placebo-controlled 3-arm parallel group trial whether optimal programming versus standard rate-response programming versus no rate-response programming for 6 months leads to appreciable improvements in exercise time and quality of life, while having no adverse effects on left ventricular function and battery longevity and what the mechanisms of this might be.

450 patients with CHF and a pacemaker will undergo the non-invasive echocardiographic assessment to establish the force frequency relationship and the optimal heart rate for contractility. They will then perform a treadmill walk test, complete quality of life questionnaires and be offered the opportunity to participate in a series of mechanistic substudies. They will then be randomised to optimal rate-response settings, standard rate response settings or no rate-response settings and followed up at 6 months at which point the tests will be repeated.

DETAILED DESCRIPTION:
Detailed Description:

Design: This will be a randomised, double-blind 'placebo' controlled trial of optimised programming versus standard rate-response settings, aiming to determine whether the short term improvements translate into longer term benefits.

Study participants: 450 adult patients (>18years).

Study Procedures: Patients attending the heart failure clinic, the pacemaker clinic or previous research participants will be approached with a standard letter and information sheet and then a telephone call to make sure any remaining questions are answered.

Patients agreeing to participate will attend the clinical research facility (CRF) and will be asked to sign a consent form. Each patient will have a standard device check, check of their demographic data, and co-morbidities. The investigators will record a resting cardiac ultrasound, and measure the force frequency relationship (FFR) to determine critical heart rate (HR), and the optimal range of HR rise. All images will be stored for offline analysis. Participants will then be asked to do a symptom-limited walk test on the treadmill (until they cannot do any more). At this first visit, participants will also complete quality of life questionnaires and be invited to participate in substudies including cardiac magnetic resonance, blood tests, tests of autonomic dysfunction. All of these activities will take place in the Clinical Research Facility at Leeds General Infirmary.

Randomisation: Each patient will then be randomised to either optimised programming (n=225) as predicted by their force-frequency curve (n=200), standard settings (n=112) or no rate response programming (n=113). In the optimised group, programming will keep heart rates below the critical HR. Randomisation will be by a random number generator and programming will be undertaken by one of my colleagues to maintain blinding.

Follow-up: Each patient will be called at one month to check that they are tolerating any changes and will then be invited back at 6 months for a repeat resting echocardiogram, treadmill walk test and quality of life assessment.

Data: All data will be stored on a bespoke Excel spreadsheet on an LTHT server in a password-protected folder.

Primary Endpoint: The effects of heart rate programming that optimises heart rate for contractility on change in treadmill-based walk distance over six months in patients with heart failure and a pacemaker.

Secondary endpoints: 1) the safety of pacemaker programming optimised for heart rate in patients with heart failure and a pacemaker, 2) the effect of this programming on change of quality of life at 6 months 3) the effect of this programming on change in cardiac function at 6 months.

Mechanistic endpoints: 1) The effect of heart rate programming on measures of autonomic function, 2) Changes in cardiac function during exercise, 3) The effect of optimised heart rate programming on strain, wall stress and perfusion by cardiac magnetic resonance, 4) changes in biomarkers associated with heart failure

ELIGIBILITY:
Inclusion Criteria:

* Clinical, echocardiographic and neurohormonal evidence of heart failure
* Cardiac pacemaker,
* Able to perform a peak exercise test,
* Willing and able to give informed consent.

Exclusion Criteria:

* Angina pectoris symptoms limiting exercise tolerance,
* Unstable heart failure symptoms (medical therapy changes in last three months), Poor image quality,
* Calcium channel blockers (CCBs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Treadmill walk time | 6 months
  Time walked during a standard incremental treadmill test

SECONDARY OUTCOMES:
Quality of life 1 | 6 months
  EQ5D-5L score
Quality of life 2 | 6 months
  KCCQ score
Clinical composite score | 6 months
  Clinical outcomes combined (death, hospitalisation, NYHA symptom level, diuretic dose
Cardiac function during exercise measured by LVEF on echocardiogrpahy | 6 months
  As assessed on a cycle ergometer
Wall stress by cardiac MRI | 6 months
  Wall stress assessed by cardiac MRI
Autonomic dysfunction | 6 months
  Measures of Muscle Sympathetic Nerve Activity
Autonomic dysfunction | 6 months
  Heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: John Gierula, PhD, Principal Investigator — University of Leeds
Locations (1):
- Leeds General Infirmary, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An application with appropriate ethical approval is made to the corresponding author and the deidentified data would be transferred securely to servers of the applicant's organisation.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after initial analysis and within three months of an apporoved request being made.
Access Criteria: A request is made that the applicant's organisation deem ethically justified, and for which ethical approval is in place, and an analysis plan is available.